CLINICAL TRIAL: NCT00703079
Title: Impact of Somatostatin Analogs vs. Surgery on Glucose Metabolism in Acromegaly: Results of a 5 Years Observational, Open, Prospective Study
Brief Title: Impact of Somatostatin Analogs vs. Surgery on Glucose Metabolism in Acromegaly
Acronym: GLUSSA
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Annamaria Colao, Department of Molecular and Clinical Endocrinology and Oncology
Other Study IDs: NeuroendoUnit-10
Record Dates: First submitted 2008-06-20; First posted 2008-06-23 (Estimated); Last update posted 2008-06-23 (Estimated); Status verified 2008-06

CONDITIONS: Acromegaly
Keywords: Acromegaly; GH; IGF-I; Octreotide-LAR; Lanreotide; Transsphenoidal surgery
MeSH Terms: conditions — Acromegaly | interventions — lanreotide; lactitol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Sera from most patients on a yearly bases are stored in our freezed at minus 80° for eventual further studies. No experimental parameters are included in the current study.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Group A: >15 patients treated only with SSA (octreotide-LAR or lanreotide depot)
  Interventions: Drug: Octreotide-LAR or lanreotide
- Group B: >15 patients treated with surgery after a period of SSA treatment of 6-24 months
  Interventions: Drug: Octreotide-LAR or lanreotide; Procedure: Transsphenoidal adenomectomy
- Group C: >15 patients cured after surgery only
  Interventions: Procedure: Transsphenoidal adenomectomy
- Group D: >15 patients treated with surgery first and then with SSA after 6-12 months
  Interventions: Drug: Octreotide-LAR or lanreotide; Procedure: Transsphenoidal adenomectomy

INTERVENTIONS:
Drug: Octreotide-LAR or lanreotide — Treated with octreotide-LAR will be given at dosages of 10-40 mg/q28d and treatment with lanreotide-SR at dosages of 60-120 mg/q28d. The dosages are up-titrated to control GH and IGF-I levels
  Other Names: Sandostatin-LAR (Novartis), Ipstyl (Ipsen)
  Groups: Group A; Group B; Group D
Procedure: Transsphenoidal adenomectomy — Removal of pituitary adenomas via one-nostril transsphenoidal approach and endoscopy-assisted.
  Groups: Group B; Group C; Group D

SUMMARY:
To investigate the 60 month impact of surgery and somatostatin analogues (SSA) on glucose metabolism in acromegaly we will analyzed data from 100 patients with acromegaly according with different treatments (group A=with SSA only; group B= SSA followed by surgery; group C= surgery only; group D= surgery followed by SSA). At diagnosis and after 6-12 and 60 months were analyzed as primary outcome measure changes in fasting glucose and as secondary outcome measures changes of glycated hemoglobin (HbA1c) and insulin levels, HOMA-R and HOMA-β, representing insulin resistance and β-cell function, respectively.

We will enrol 100 patients and expect half of them to have IGT or diabetes mellitus. We do not expect changes according with different treatment after 60 months while SSA-treated patients might experience deterioration of glucose tolerance after 6-12 months. We intend to look for predictors of deterioration of glucose tolerance.

DETAILED DESCRIPTION:
Impaired glucose tolerance (IGT) and overt diabetes mellitus are frequently associated with acromegaly. Patients with acromegaly are insulin resistant both in the liver and in the periphery, displaying hyperinsulinemia and increased glucose turn-over in the basal post-absorptive states. The prevalence of diabetes mellitus and that of IGT in acromegaly is unknown but is reported to range 19-56% and 16-46% in different series. The increased cardiovascular morbidity and mortality associated with acromegaly may party be a consequence of the increased insulin resistance that frequently accompanies GH excess. Glucose tolerance may worsen in patients treated with somatostatin analogues (SSA), because insulin secretion, i.e. β-cell function, is also suppressed. SSA induce control of GH and IGF-I excess in approximately 60% of patients after 12 months of treatment with no significant difference as applied after unsuccessful surgery or as first-line in newly diagnosed patients and control of GH and IGF-I levels occur with an even higher prevalence after a longer period of treatment. The inhibitory effect of SSA on pancreatic insulin secretion might, however, complicate the overall effect of this treatment on glucose tolerance. We recently demonstrated that 12 months after first-line treatment with SSA or surgery produced a similar improvement in LV hypertrophy and diastolic filling while systolic function increased more evidently in SSA-treated patients, total/HDL-cholesterol ratio significantly reduced only in SSA-treated patients while fasting glucose levels significantly reduced only in surgery-treated patients. A normal pituitary function was found in 46.4% of SSA-treated and in 36.4% of surgery-treated patients, resulting unchanged in the former and slightly reduced in the latter. Both a direct effect of SSA and a more preserved pituitary function might explain these results. Longitudinal data of glucose tolerance in patients with acromegaly and with or without diabetes treated long-term with SSA or surgery or both are still very limited.

In order to investigate whether SSA negatively impact glucose tolerance in acromegaly, we will analyze data collected prospectively during a 10 year period. We will compare the results of glucose tolerance at diagnosis after 6-12 months and after 60 months of treatment with SSA or surgery. Patients will be grouped according with their treatment (SSA only, surgery only, SSA followed by surgery and SSA followed by surgery and SSA) in order to establish the effects on glucose tolerance mediated by disease control and type of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with either first-line surgery via trans-sphenoidal route by microscopic and/or endoscopic approach or with first-line depot SSA treatment, or both and
* Patients with available follow-up after 60 months of treatment

Exclusion Criteria:

* Patients requiring dopamine-agonists or pegvisomant
* Patients receiving the s.c. octreotide for longer than 15 days
* Patients receiving radiotherapy,
* Patients with a follow-up shorter than 60 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will review all files from consecutive patients with active acromegaly coming to the Units of Endocrinology or Neurosurgery of the "Federico II" University of Naples from Jan 1st 1997 to June 1st 2008, primarily treated with either surgery or depot SSA, i.e. lanreotide (LAN) or slow-release octreotide (LAR), and with an available follow-up of at least 60 months. Due to the study design, this is a non ran-domized study. However, our routine procedure generally considers first-line treatment with SSA for 6-12 months, unless the tumors are clearly non invasive on Magnetic Resonance Imaging (MRI) and/or the patients who do not present any surgical or anesthesiological risk.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 1997-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Changes of fasting glucose levels. | 0, 6-12 and 60 months

SECONDARY OUTCOMES:
changes in Hb1Ac levels changes in fasting insulin levels changes in HOMA-R index changes in HOMA-β index | 0, 6-12, 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Annamaria Colao, MD, Principal Investigator — Federico II University
Locations (1):
- Department of Molecular and Clinical Endocrinology and Oncology, University Federico II of Naples, Naples, Italy

REFERENCES:
- [Result] Colao A, Ferone D, Marzullo P, Lombardi G. Systemic complications of acromegaly: epidemiology, pathogenesis, and management. Endocr Rev. 2004 Feb;25(1):102-52. doi: 10.1210/er.2002-0022. PMID 14769829
- [Result] Pereira AM, Biermasz NR, Roelfsema F, Romijn JA. Pharmacologic therapies for acromegaly: a review of their effects on glucose metabolism and insulin resistance. Treat Endocrinol. 2005;4(1):43-53. doi: 10.2165/00024677-200504010-00005. PMID 15649100
- [Result] Kasayama S, Otsuki M, Takagi M, Saito H, Sumitani S, Kouhara H, Koga M, Saitoh Y, Ohnishi T, Arita N. Impaired beta-cell function in the presence of reduced insulin sensitivity determines glucose tolerance status in acromegalic patients. Clin Endocrinol (Oxf). 2000 May;52(5):549-55. doi: 10.1046/j.1365-2265.2000.00986.x. PMID 10792333
- [Result] Lamberts SW, Uitterlinden P, Verschoor L, van Dongen KJ, del Pozo E. Long-term treatment of acromegaly with the somatostatin analogue SMS 201-995. N Engl J Med. 1985 Dec 19;313(25):1576-80. doi: 10.1056/NEJM198512193132504. PMID 2866445
- [Result] Colao A, Pivonello R, Galderisi M, Cappabianca P, Auriemma RS, Galdiero M, Cavallo LM, Esposito F, Lombardi G. Impact of treating acromegaly first with surgery or somatostatin analogs on cardiomyopathy. J Clin Endocrinol Metab. 2008 Jul;93(7):2639-46. doi: 10.1210/jc.2008-0299. Epub 2008 Apr 29. PMID 18445662
- [Result] Colao A, Pivonello R, Auriemma RS, Galdiero M, Savastano S, Lombardi G. Beneficial effect of dose escalation of octreotide-LAR as first-line therapy in patients with acromegaly. Eur J Endocrinol. 2007 Nov;157(5):579-87. doi: 10.1530/EJE-07-0383. PMID 17984237
- [Result] Colao A, Martino E, Cappabianca P, Cozzi R, Scanarini M, Ghigo E; A.L.I.C.E. Study Group. First-line therapy of acromegaly: a statement of the A.L.I.C.E. (Acromegaly primary medical treatment Learning and Improvement with Continuous Medical Education) Study Group. J Endocrinol Invest. 2006 Dec;29(11):1017-20. doi: 10.1007/BF03349217. No abstract available. PMID 17259801
- [Derived] Colao A, Auriemma RS, Galdiero M, Cappabianca P, Cavallo LM, Esposito F, Grasso LF, Lombardi G, Pivonello R. Impact of somatostatin analogs versus surgery on glucose metabolism in acromegaly: results of a 5-year observational, open, prospective study. J Clin Endocrinol Metab. 2009 Feb;94(2):528-37. doi: 10.1210/jc.2008-1546. Epub 2008 Nov 11. PMID 19001517